CLINICAL TRIAL: NCT01438502
Title: "The Impact of Hypertonic Saline/ Colloids Infusion During Cardio-pulmonary-bypass in Patients Expected Long CPB-time"
Brief Title: "The Effect of Reduced Fluid Load After Cardiac Surgery"
Status: Withdrawn | Type: Observational
Why Stopped: Changes in staff resulted in logistic difficulties to perform the study
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/491
Record Dates: First submitted 2011-09-19; First posted 2011-09-22 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Fluid Overload; Organ Edema; Organ Function
Keywords: cardiac surgery; cardio-pulmonary-bypass
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HyperHAES
  Interventions: Drug: HyperHAES® (hypertonic saline/HES)

INTERVENTIONS:
Drug: HyperHAES® (hypertonic saline/HES) — After arrival to the operating theatre both study groups will receive an infusion of acetated Ringers solution 4 ml/kg/hour. Additionally both groups for 4 hours will receive 1 ml/kg/hour of a blinded solution. This solution will be either acetated Ringers solution or HyperHAES® (7.2 % NaCl/ 6 % hydroxyethyl-starch (200/0.5)).
  Other Names: HyperHAES® (7.2 % NaCl/ 6 % hydroxyethyl-stivelse (200/0.5)

SUMMARY:
The purpose of this study is to verify that an infusion of hypertonic saline/colloids during cardio-pulmonary-bypass will reduce fluid overload and organ edema for cardiac patients with expected long-CPB-time.

Expected beneficial effects are improved organ function for heart and lungs.

DETAILED DESCRIPTION:
Fluid overloading with oedema formation is a regular finding following on-pump cardiac surgery and may contribute to postoperative organ dysfunction. Myocardial oedema has been reported to impair both systolic and diastolic function. An association between intraoperative fluid loading and postoperative adverse outcome has been demonstrated in cardiac patients.

Our group has experience with the use of hypertonic saline/colloids in several experimental studies (pigs). In these animal studies we have used hypertonic saline/colloids both as an infusion during CPB or as an additive to CPB-prime. Both administration methods resulted in significant reduction in fluid loading due to better intravascular volume preservation.

One clinical study from our group observed reduced fluid load and an improved cardiac index when an infusion of hypertonic saline/colloids was used during cardiac surgery. Patients included in this study had a normal left ventricular function and no co-morbidity.

The planned study includes patients with combination procedures, both aorta coronary bypass and valve implantation, and expected long CPB-time.Time spent on CPB is a individual risk factor negatively associated with increased mortality and morbidity. The investigators believe high-risk patients will have even more benefit of reduced fluid loading. Their tolerance for hypovolemia is lower and the incidence for hemodynamic instability first hours postoperatively is greater.

The patients will be randomized to receive either a continuous infusion of hypertonic saline/colloids or acetated Ringer's solution during CPB. Accurate accounts of fluid additions, blood loss and diuresis will be kept. Determination of cardiac output (C.O.), intrathoracic blood volume (ITBV), extravascular lung water (EVLW) and global end diastolic volume (GEDV) will be monitored by use of the transpulmonary thermodilution technique PiCCO®plus system.

Preoperative and postoperative echo cor will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for combination surgery, both elective coronary bypass and valve surgery, with expected long CPB-time, and who after orally and written information agrees to participate in the study.

Exclusion Criteria:

* Age less than 18 years
* Serum-Sodium higher than 145 mmol/l
* Hematocrit less than 30 %
* Estimated GFR less than 60
* BMI more than 30 or BMI less than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Reduction of organ edema and improved organ function | 24-hours postoperatively
  As a target for effect the investigators have chosen to study improvements for organ function. Indexed values for cardiac output (CI) measured by the PICCO system will be a parameter for heart function, and lung function will be measured by EVLWI (extravascular lung water index), paO2/FiO2 -ratio and time spent in respirator. Additionally a strict account for fluid balance will be kept.